CLINICAL TRIAL: NCT00968487
Title: A Clinical Study of the Safety of Ascending Doses of Autologous Lyophilized Plasma Versus Fresh Frozen Plasma in Normal Healthy Volunteers
Brief Title: The Safety of Autologous Lyophilized Plasma Versus Fresh Frozen Plasma in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-I-LyP-1
Record Dates: First submitted 2009-08-26; First posted 2009-08-31 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Lyophilized Plasma; Fresh Frozen Plasma; Hemorrhage; Coagulopathy; Autologous; HemCon; Plasmapheresis; Freeze Drying; Transfusion; Resuscitation; Safety of Lyophilized Plasma in Normal, Healthy Volunteers
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lyophilized Plasma (Experimental)
  Interventions: Biological: Lyophilized Plasma
- Fresh Frozen Plasma (Active Comparator)
  Interventions: Other: Fresh Frozen Plasma

INTERVENTIONS:
Biological: Lyophilized Plasma — Lyophilized Plasma is serves as a source of plasma proteins for subjects who are deficient in plasma proteins. The donor and recipient are the same person, therefore the process is autologous. HemCon's lyophilized plasma originates from FFP from screened individual donors to significantly reduce the risk of bloodborne disease transmission and undesired transfusion-associated reactions. Each single-donor unit is tested (per required of the blood supply) to reduce the risk of transmission of infectious agents and hence, maximize subject safety.
  Arms: Lyophilized Plasma
Other: Fresh Frozen Plasma — The fluid portion of one unit of human blood that has been centrifuged, separated, and frozen solid at -18 °C (-0.4 °F) (or colder) within 6 hours of collection.
  Arms: Fresh Frozen Plasma

SUMMARY:
A single-site, single-blind study of ascending doses of Lyophilized Plasma in normal healthy volunteers.

DETAILED DESCRIPTION:
This "first-in-human" Phase I, single-center, dose escalation study (using 3 dose levels) is proposed to assess the safety of infusing reconstituted lyophilized human plasma (LyP). The study design incorporates plasmapheresis-derived autologous plasma (FFP) for infusion(s) to eliminate variables and events known to be related to allogenic transfusion. Subjects will be enrolled at a blood center and provide autologous FFP that will be shipped to the sponsor site and used as the starting material to manufacture LyP. Once manufacturing is complete, the LyP (autologous) will be returned to the blood center for reconstitution and infusion into subjects. Maximum dosage within this study will approach "massive transfusion" (1 liter in Cohort 3) to obtain a preliminary assessment of safety. One half of the FFP obtained from subjects in Cohort 3 (only) will be shipped to the sponsor and returned to the site (but not manufactured into LyP) to serve as the control (autologous FFP).

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant/ non-breast feeding females as they present interest
* Minimum weight, 140 pounds (64 kg) or 175 pounds for Cohort 3 only
* Ages 18-55 years
* Subject self-reports that he/she feels well and healthy
* Subject is able to donate one unit of whole blood based on the AABB donor history questionnaire with modifications indicated. Volunteers with history of travel which puts them at risk for vCJD will be eligible to participate.
* Has read the educational materials on donating blood and has had his/her questions answered
* Able and willing to provide informed consent
* Available for the duration of the trial (approximately 8 weeks for Cohorts 1 and 2 and 12 weeks for Cohort 3) and able to come to the treatment clinic for scheduled study visits.
* Females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective medically accepted contraceptive regimen. A highly effective method of birth control is defined as those which result in a lower failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner.
* Female subjects must have a negative serum pregnancy test prior to enrollment.
* Understands the English language
* Scored greater or equal to 35 on the Duke Activity Status Index (DSAI)

Exclusion Criteria:

* Known liver, kidney, cardiovascular, neurologic, gastrointestinal, blood, endocrine/ metabolic, autoimmune or pulmonary disease; treated or untreated hypertension (see precise cut-off below)
* Cancer of any kind, under treatment or resolved
* Known or past coagulopathy conditions or blood disease
* Currently using medications for anticoagulant therapy
* Currently taking fish oil supplements
* Any conditions, medications, etc. on the AABB medical deferral list
* Previous use of clotting factor concentrate(s)
* Past diagnosis of stroke or transient ischemic attack
* Current or history of drug or alcohol abuse. Used needles to take drugs, steroids, or anything not prescribed by a doctor
* Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness or received a positive test result for HIV infection.
* Current or past infection with Hepatitis B or Hepatitis C virus
* Has received positive test for Syphilis
* Has received positive test for West Nile Virus
* Female subject who is pregnant, lactating or with a positive pregnancy test
* Currently taking an antibiotic or another medication for an infection.
* Treatment or use of aspirin (or other platelet inhibiting agents) within 14 days of study donation and infusion visits
* In the past week, has had a headache and fever at the same time.
* Known intolerance to citric acid.
* Receipt of blood or blood products within the past 12 months
* Systolic blood pressure greater than 180 mmHg
* Diastolic blood pressure greater than 90 mmHg
* Temperature greater than 100° F
* Hematocrit will not be less than 38% for both male and female donors
* History of current mental or psychiatric condition
* Treatment with any investigational agent within one month before treatment application for this trial
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment
* Subject is institutionalized because of legal or regulatory order
* Other criteria based upon the AABB universal donor history questionnaire with the exception of travel to a vCJD area (i.e. travel to a vCJD area is not a study exclusion).
* Has had any vaccinations or injections in the past 8 weeks.
* Is a Medicare recipient
* Is uninsured (does not have health care insurance)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of increasing doses of infused autologous units of LyP in normal healthy volunteers and to define possible LyP adverse reactions. | 1 day, 7 day, 14 day, and 28 day follow-ups after infusion.

SECONDARY OUTCOMES:
To demonstrate that coagulation function assays and specific coagulation factors [Cohort 3 only] are similar within clinically meaningful levels, post-infusion of either autologous LyP or FFP. | 1 day, 7 day, 14 day, and 28 day follow up after second infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cancelas, M.D., Ph.D., Principal Investigator — Hoxworth Blood Center
Locations (1):
- Hoxworth Blood Center, Cincinnati, Ohio, United States